CLINICAL TRIAL: NCT00384215
Title: Insulin Glargine [rDNA Origin] Injection vs Pioglitazone as add-on Therapy in Patients Failing Monotherapy With Sulfonylurea or Metformin: a Randomized, Open, Parallel Study
Brief Title: Insulin Glargine [rDNA Origin] Injection vs Pioglitazone as add-on Therapy in Patients Failing Monotherapy With Sulfonylurea or Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4020
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: insulin glargine [rDNA origin] injection

SUMMARY:
This trial will explore the various advantages and possible disadvantages of pioglitazone and insulin glargine when added to monotherapy. Glycemic control, hypoglycemia, weight, lipid profiles, quality of life and cost will be studied given a comprehensive set of data that may help future treatment decisions.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

1. Diagnosis of type 2 diabetes mellitus for at least six months
2. Continuous treatment with at least 1g metformin or half maximally labeled dose of a SU daily for at least three months
3. HbA1c >/= 8 % and </= 12%, inclusive, as measured at screening week
4. Willingness to accept, and demonstrated ability to inject insulin glargine therapy
5. Demonstrated ability and willingness to perform SMBG using a plasma-referenced glucose meter at least twice a day
6. Ability to understand and willingness to adhere to and be compliant with the study protocol

EXCLUSION CRITERIA:

1. Stroke, myocardial infarction (MI), coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) or angina pectoris within the last 12 months
2. Congestive heart failure requiring pharmacological treatment
3. Impaired renal function, as shown by but not limited to serum creatinine >/= 1.5 mg/dl (133µmol/L) for males, or >/= 1.4 mg/dl (124 µmol/L) for females
4. Treatment with non-selective beta-blockers (including ocular)
5. Acute infection
6. History of or presence of signs of significant peripheral edema
7. Acute or chronic or history of metabolic acidosis, including diabetic ketoacidosis
8. Planned radiological examinations requiring administration of contrasting agents
9. Clinical evidence of active liver disease, or serum ALT 2.5 times the upper limit of the normal range
10. History of hypoglycemia unawareness
11. Pregnant or breastfeeding females
12. Failure to use adequate contraception (women of current reproductive potential only)
13. BMI < 25 kg/(m)(m)
14. Treatment with systemic steroids or large doses of inhaled steroids
15. Treatment with any diabetes medication other than the medications required by this study
16. Use of an investigational drug within the previous month
17. Known hypersensitivity to insulin glargine, pioglitazone or any of the components of insulin glargine and pioglitazone
18. Any malignancy within the last five years, except adequately treated basal cell carcinoma and adequately treated cervical carcinoma in situ.
19. Current addiction or alcohol abuse or history of substance or alcohol abuse within two years
20. Diagnosis of dementia
21. Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with completion of the study or interpretation of study results
22. Inability to comply with study procedures

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352
Dates: Start 2001-12; Study Completion 2005-02

PRIMARY OUTCOMES:
To determine whether glycemic control as measured by HbA1c is different between insulin glargine [rDNA Origin] injection and pioglitazone when added to subjects who fail monotherapy with SU or metformin.

SECONDARY OUTCOMES:
Compare occurrence of hypoglycemia
Compare change in body weight
Compare change in FPG
Compare change in serum lipid profile
Compare percentage of subjects achieving HbA1c levels </= 7%
Compare the time until an HbA1c </= 7% is achieved
Compare change in HRQOL
Compare cost of therapy for hyperglycemia treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, B.S., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States